CLINICAL TRIAL: NCT05789810
Title: Effects of Applications Manual Pressure and ShotBlocker to Reduce Needle-Related Pain and Fear in Children With Type 1 Diabetes Mellitus
Brief Title: Manual Pressure and ShotBlocker to Reduce Needle-Related Pain and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Collaborators: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, İLKNUR GÖL, Assoc. Prof, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Çankırı Karatekin Üniversitesi
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Pain; Fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manuel pressure group (Experimental): 10-second manual pressure was applied on the insulin injection area. The injection point was pressed by the diabetes nurse's right thumb over the site until resistance was felt and the pressure was then maintained for 10 seconds before the insulin injection. Then insulin injection was administered.
  Interventions: Other: Manuel pressure
- ShotBlocker group (Experimental): ShotBlocker device was placed in the insulin injection site by contacting the protruding surface with the skin and was kept throughout the injection. The injection was applied through the opening at the middle of the tool.
  Interventions: Other: ShotBlocker
- Control group: (Experimental): No intervention was performed to reduce pain and fear.
  Interventions: Other: Control

INTERVENTIONS:
Other: Manuel pressure — 10-second manual pressure was applied on the insulin injection area.
  Arms: Manuel pressure group
Other: ShotBlocker — ShotBlocker device was placed in the insulin injection site by contacting the protruding surface with the skin and was kept throughout the injection. The injection was applied through the opening at the middle of the tool.
  Arms: ShotBlocker group
Other: Control — No intervention was performed to reduce pain and fear.
  Arms: Control group:

SUMMARY:
This experimental, prospective, and randomized controlled study was designed to determine and compare the effects of applying manual pressure and ShotBlocker methods in reducing pain and fear during the subcutaneous insulin injection for children with Type 1 diabetes mellitus. A parallel trial design was used describing two intervention (manual pressure and ShotBlocker) and a control group (no intervention used) as the third arm. The study population consisted of children aged 6-12 years, diagnosed with Type 1 diabetes mellitus, administered insulin injections, able to cognitively score their pain and fear levels, who wanted to participate in the study, and gave verbal and written consent to participate in the study.The study sample composed of 90 children based on confidence interval of 95% and statistical power of 80%. Each intervention and control group was matched in terms of gender. In the study, the randomization of the sample group was performed by using stratification and block randomization methods.

DETAILED DESCRIPTION:
This experimental, prospective, and randomized controlled study was designed to determine and compare the effects of applying manual pressure and ShotBlocker methods in reducing pain and fear during the subcutaneous insulin injection for children with Type 1 diabetes mellitus. A parallel trial design was used describing two intervention (manual pressure and ShotBlocker) and a control group (no intervention used) as the third arm. The study sample composed of 90 children based on confidence interval of 95% and statistical power of 80%. In post-hoc analysis made using G power 3.1 software, the power of sample size including 90 children with α = .05 and effect size (w)= .31, was 1 - β = 0.87. Power of .80 or higher is indicative of an adequate sample size. In addition, in order to prevent bias and increase the validity of the data, the pain and fear scores of the children before and after the procedure were assessed by three different groups as children (n:90), their parents (n:90), and a researcher specialized in pediatric nursing (the first author; n:1), and the inter-observer agreement was examined. The parents meeting the following inclusion criteria were eligible for the participation: 1) being healthy in terms of neurological functions, 2) communicating verbally, 3) understanding and reading Turkish, and 4) voluntarily signing the written informed consent. The children were first categorized according to their genders and then assigned into three study groups by using block randomization method to control the effect of gender on pain. First, the numbers 1, 2 and 3, representing the three groups, were written on paper of the same color and shape and put in a pink box for girls and blue for boys.After, female children were asked to draw a piece of paper from the pink box and male children were asked to draw a piece of paper from the blue box to provide a randomized distribution and to reduce all negative effects. Thus, the groups became self-balanced. Intervention and control groups were matched in themselves based on gender, each group included a total of 30 children including 15 girls and 15 boys. The study was conducted in accordance with the CONSORT guideline for reporting the randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

administered insulin injection, able to score cognitively pain and fear levels, who want to participate in research children who gave verbal and written consent to participate in the study

Exclusion Criteria:Having pacemaker and neurodevelopmental disorder, having lipodystrophy, infection and nerve damage in the injection area, administered analgesics in the last 6 hours, admitted to the outpatient clinic with a picture of ketoacidosis, Diagnosed with Reynaud's syndrome and sickle cell anemia children who do not want to participate in the research

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 5 Months
  Wong-Baker FACES Pain Rating Scale was used to assess the pain levels of children before and after the insulin administration. This scale was administered to the children, their parents, and a researcher (the first author) within 5 minutes before and immediately after the insulin administration. The scale was scored blindly before and after the insulin administration so that they were not affected by each other.
Fear Severity | 5 Months
  Child Fear Scale was used to assess pain-related fear levels of children before and after the insulin administration. This scale was administered to the children, their parents, and a researcher (the first author) within 5 minutes before and immediately after the insulin administration. The scale was scored blindly before and after the insulin administration so that they were not affected by each other.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin Univesity, Çankiri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girgin BA, Gol I, Gozen D, Carikci F, Kirmizibekmez H. Effects of applications manual pressure and shotblocker to reduce needle-related pain and fear in children with type 1 diabetes mellitus. J Pediatr Nurs. 2023 Nov-Dec;73:84-90. doi: 10.1016/j.pedn.2023.08.024. Epub 2023 Aug 30. PMID 37651942